CLINICAL TRIAL: NCT06650137
Title: Evaluation of the Relevance of Diaphragmatic Stroke Ultrasound for the Etiological Diagnosis of Acute Respiratory Distress in an Emergency Department: a Prospective Multicenter Study.
Brief Title: Evaluation of the Relevance of Diaphragmatic Stroke Ultrasound for the Etiological Diagnosis of Acute Respiratory Distress in an Emergency Department.
Acronym: EchoDiaph
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL23_0425
Record Dates: First submitted 2024-10-04; First posted 2024-10-21 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Pneumonia; Diaphragm; Movement; Diaphragmatic Ultrasound; Emergency Medical Services; Acute Respiratory Distress Syndrome (ARDS)
Keywords: Diaphragmatic ultrasound,; ultrasonography; Pneumonia; Diaphragm; Acute respiratory failure; Emergency; Diaphragmatic excursion
MeSH Terms: conditions — Pneumonia; Respiratory Distress Syndrome; Emergencies

STUDY DESIGN:
Intervention Model Description: Prospective interventional multicenter diagnostic study
Masking Description: The reference will be the etiological diagnosis based on expert opinion. Two experts (physicians experienced in the management of ARD) will judge, blind to each other and to the judgement criteria, the cause of the ARD on the basis of a medical file review at least one month after the ARD episode.
  Ultrasound measurements will be analyzed a posteriori by an investigator blind to the results of the gold standard.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adult emergency patients with acute respiratory distress (Experimental): Subjects aged ≥ 18 years presenting to the emergency department with ARD defined by respiratory rate (RR) > 25 and/or signs of struggle.
  Every potentially eligible patient will have a right diaphragmatic ultrasound performed by a doctor trained in the technique.
  Interventions: Diagnostic Test: diaphragmatic ultrasound

INTERVENTIONS:
Diagnostic Test: diaphragmatic ultrasound — The examination is performed with a phased array probe, also known as a cardiac probe. The technique used will be that described and validated in anterior studies: the patient is in the Fowler position: half-seated, at an angle of around 45 degrees. The patient is ventilating spontaneously, and no participation is required. The probe is positioned in the sub-costal region between the mid-clavicular and anterior axillary line on the right, and between the anterior and middle axillary line in the sub- or intercostal region on the left. The liver is used as an acoustic window for the right hemi-diaphragm. The probe is oriented medially, cranially and dorsally.
  The operator switches to time-motion (TM) mode when an angle of over 70° is achieved between the upper part of the diaphragm and the analysis axis in the most cephalic part of the diaphragm. The image is frozen when 6 respiratory cycles have been measured.

SUMMARY:
The goal of this Prospective interventional multicenter diagnostic study is to investigate the use of diaphragmatic ultrasound (DE) as a diagnostic tool in an adult emergency department for patients in acute respiratory distress.

The main question it aims to answer is to evaluate the relevance of measuring the Sum of Plateau Times (SPT) by Clinical Ultrasound in Emergency Medicine (CHEM) for the diagnosis of pneumopathy during acute respiratory distress (ARD) in the Emergency Department.

Secondary objectives include the study of other diaphragmatic ultrasound parameters, inspiratory plateau time (IPT) and expiratory plateau time (EPT), and the diagnostic relevance of PTS for the diagnosis of decompensation of Chronic obstructive pulmonary disease (BPCO) and acute cardiogenic pulmonary edema (APO).

Each eligible patient will have a right diaphragmatic ultrasound performed by a trained physician, then clinicobiological data will be collected later from medical records, and the etiological diagnosis will be established by a committee of 2 experts in the management of respiratory distress.

DETAILED DESCRIPTION:
Diaphragmatic ultrasound (DE) has never been studied as a diagnostic tool in the emergency department. The sensitivity and specificity of pleural ultrasound for the diagnosis of pneumopathy is superior to that of chest radiography, with evidence of interstitial syndrome or unilateral pleural effusion, but it is not specific for infectious pneumopathy. Proving that diaphragmatic ultrasonography can be used to diagnose pneumopathy in respiratory distress, thanks to a specific index known as the Sum of Plateau Times (STP), will save time in patient management.

The secondary criteria of this study could be used in future studies, if they prove relevant.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older;
* Patient with ARD defined by respiratory rate (RR) strictly superior to 25 and/or signs of struggle which are: thoraco-abdominal rocking, active abdominal breathing, recruitment of extra-diaphragmatic respiratory muscles AND
* peripheral saturation (SpO2) strictly inferior to 90% and/or hypercapnic acidosis (pH strictly inferior to 7.35 and pCO2 strictly superior to 45mmHg) on arterial blood gases;
* Spontaneous ventilation.
* Patients presenting a clinical severity score of Grade 1 with signs of struggle, as well as those with Grade 2 and Grade 3. A clinical severity score will be used as follows: Grade 1: Minimal polypnoea with respiratory rate (RR) between 20 and 25 ; Grade 2: Moderate polypnoea with respiratory rate (RR) between 25 and 35; Grade 3: Major polypnoea with respiratory rate (RR) between 35 to 50.

Exclusion Criteria:

* Adult protected by law (guardianship, curatorship, legal protection)
* Refusal of consent after information
* Patient on non-invasive ventilation ;
* Patient on mechanical ventilation;
* Respiratory rate superior to 50/min
* Patient currently being treated for infectious pneumopathy with antibiotics;
* Pregnant or breast-feeding women;
* Patients with any known history of diaphragmatic pathologies.
* Illiterate or unable to understand the purpose and methodology of the study.
* Patient not affiliated to a social security scheme or not benefiting from such a scheme.
* Person deprived of liberty (by judicial or administrative decision, or forced hospitalization)
* Person participating in another study with an exclusion period still in progress,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Assess the relevance of Sum of plateau times (STP) measurement by diaphragmatic ultrasound for the diagnosis of pneumopathy during acute respiratory distress (ARD) in an emergency department. (Specificity) | Baseline
  STP (in seconds) is a sum of inspiratory plateau time (IPT) and expiratory plateau time (TPE) measured in seconds.
  TPE is defined as the time between the end of diaphragmatic descent and the start of its ascent, measured by recording Diaphragmatic curves (DC).
  TPI is defined as the time between the end of diaphragmatic ascent and the start of its descent.
  These measurements will be carried out after the ultrasound on the diaphragmatic movements recorded.
  The diagnosis will be established on the basis of medical records by two independent experts.
  intrinsic diagnostic performance will be analyzed by specificity in percentage.
  specificity corresponds to the probability of STP of giving a negative diagnosis of pneumopathy among participants without pneumopathy according to expert review of medical records (gold standard)
Assess the relevance of Sum of plateau times (STP) measurement by diaphragmatic ultrasound for the diagnosis of pneumopathy during acute respiratory distress (ARD) in an emergency department. (sensibility) | Baseline
  STP (in seconds) is a sum of inspiratory plateau time (IPT) and expiratory plateau time (TPE) measured in seconds.
  TPE is defined as the time between the end of diaphragmatic descent and the start of its ascent, measured by recording Diaphragmatic curves (DC).
  TPI is defined as the time between the end of diaphragmatic ascent and the start of its descent.
  These measurements will be carried out after the ultrasound on the diaphragmatic movements recorded.
  The diagnosis will be established on the basis of medical records by two independent experts.
  intrinsic diagnostic performance will be analyzed by sensibility in percentage.
  sensitivity corresponds to the probability of STP of giving a positive diagnosis of pneumopathy among participants with pneumopathy based on expert review of medical records (gold standard).
Assess the relevance of Sum of plateau times (STP) measurement by diaphragmatic ultrasound for the diagnosis of pneumopathy during acute respiratory distress (ARD) in an emergency department. (Positive predictive values) | Baseline
  STP is a sum of inspiratory plateau time (IPT) and expiratory plateau time (TPE) measured in seconds.
  TPE is defined as the time between the end of diaphragmatic descent and the start of its ascent, measured by recording Diaphragmatic curves (DC).
  TPI is defined as the time between the end of diaphragmatic ascent and the start of its descent.
  These measurements will be carried out after the ultrasound on the diaphragmatic movements recorded.
  The diagnosis will be established on the basis of medical records by two independent experts.
  Extrinsic diagnostic performance will be analyzed by Positive predictive values (PPV) in percentage.
  PPV corresponds to the probability of having pneumopathy if the PTS detects pneumopathy among participants with pneumopathy according to expert review of medical records (gold standard).
Assess the relevance of Sum of plateau times (STP) measurement by diaphragmatic ultrasound for the diagnosis of pneumopathy during acute respiratory distress (ARD) in an emergency department. (Negative predictive values) | Baseline
  STP is a sum of inspiratory plateau time (IPT) and expiratory plateau time (TPE) measured in seconds.
  TPE is defined as the time between the end of diaphragmatic descent and the start of its ascent, measured by recording Diaphragmatic curves (DC).
  TPI is defined as the time between the end of diaphragmatic ascent and the start of its descent.
  These measurements will be carried out after the ultrasound on the diaphragmatic movements recorded.
  Extrinsic diagnostic performance will be analyzed by Negative predictive values (NPV) in percentage.
  NPV corresponds to the probability of not having pneumopathy if the PTS does not detect pneumopathy among participants without pneumopathy according to the expert review of medical records (gold standard).
Assess the relevance of Sum of plateau times (STP) measurement by diaphragmatic ultrasound for the diagnosis of pneumopathy during acute respiratory distress (ARD) in an emergency department. (Positive likelihood ratio) | Baseline
  STP is a sum of inspiratory plateau time (IPT) and expiratory plateau time (TPE) measured in seconds.
  TPE is defined as the time between the end of diaphragmatic descent and the start of its ascent, measured by recording Diaphragmatic curves (DC).
  TPI is defined as the time between the end of diaphragmatic ascent and the start of its descent.
  These measurements will be carried out after the ultrasound on the diaphragmatic movements recorded.
  The diagnosis will be established on the basis of medical records by two independent experts.
  Extrinsic diagnostic performance will be analyzed by Positive likelihood ratio (PLR) in percentage. it is the ratio of true positives to false positives
Assess the relevance of Sum of plateau times (STP) measurement by diaphragmatic ultrasound for the diagnosis of pneumopathy during acute respiratory distress (ARD) in an emergency department. (Negative likelihood ratio) | Baseline
  STP is a sum of inspiratory plateau time (IPT) and expiratory plateau time (TPE) measured in seconds.
  TPE is defined as the time between the end of diaphragmatic descent and the start of its ascent, measured by recording Diaphragmatic curves (DC).
  TPI is defined as the time between the end of diaphragmatic ascent and the start of its descent.
  These measurements will be carried out after the ultrasound on the diaphragmatic movements recorded.
  Extrinsic diagnostic performance will be analyzed by Negative likelihood ratio (PLR) in percentage. It is the ratio of false negatives to true negatives

SECONDARY OUTCOMES:
Assess the relevance of the TPE for the etiological diagnosis of pneumopathy in patients managed for ARD in the emergency department. (Sensibility) | Baseline
  Sensibility %
Assess the relevance of the TPE for the etiological diagnosis of pneumopathy in patients managed for ARD in the emergency department. (Specificity) | Baseline
  Specificity %
Assess the relevance of the TPE for the etiological diagnosis of pneumopathy in patients managed for ARD in the emergency department. (Positive predictive values (%)) | Baseline
  Positive predictive values (%)
Assess the relevance of the TPE for the etiological diagnosis of pneumopathy in patients managed for ARD in the emergency department. (Negative predictive values (%)) | Baseline
  Negative predictive values (%)
Assess the relevance of the TPE for the etiological diagnosis of pneumopathy in patients managed for ARD in the emergency department. (Positive likelihood ratio (%)) | Baseline
  Positive likelihood ratio (%)
Assess the relevance of the TPE for the etiological diagnosis of pneumopathy in patients managed for ARD in the emergency department. (Negative likelihood ratio (%)) | Baseline
  Negative likelihood ratio (%)
Assessing the relevance of IPT for the etiological diagnosis of pneumopathy in patients managed for ARD in the emergency department (Sensibility ) | Baseline
  Sensibility %
Assessing the relevance of IPT for the etiological diagnosis of pneumopathy in patients managed for ARD in the emergency departmentSpecificity | Baseline
  Specificity %
Assessing the relevance of IPT for the etiological diagnosis of pneumopathy in patients managed for ARD in the emergency department. Negative predictive values | Baseline
  Negative predictive values %
Assessing the relevance of IPT for the etiological diagnosis of pneumopathy in patients managed for ARD in the emergency department. Positive likelihood ratio | Baseline
  Positive likelihood ratio %
Assessing the relevance of IPT for the etiological diagnosis of pneumopathy in patients managed for ARD in the emergency department. Negative likelihood ratio | Baseline
  Negative likelihood ratio %
Assess the relevance of PTS for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Sensibility | Baseline
  Sensibility %
Assess the relevance of PTS for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Specificity | Baseline
  Specificity %
Assess the relevance of PTS for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Positive predictive values | Baseline
  Positive predictive values %
Assess the relevance of PTS for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Negative predictive values | Baseline
  Negative predictive values %
Assess the relevance of PTS for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Positive likelihood ratio | Baseline
  Positive likelihood ratio %
Assess the relevance of PTS for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Negative likelihood ratio | Baseline
  Negative likelihood ratio %
Assess the relevance of IPT for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Sensibility | Baseline
  Sensibility %
Assess the relevance of IPT for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Specificity | Baseline
  Specificity %
Assess the relevance of IPT for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Positive predictive values | Baseline
  Positive predictive values %
Assess the relevance of IPT for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Negative predictive values | Baseline
  Negative predictive values %
Assess the relevance of IPT for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Positive likelihood ratio | Baseline
  Positive likelihood ratio %
Assess the relevance of IPT for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Negative likelihood ratio | Baseline
  Negative likelihood ratio %
Assess the relevance of TPE for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Sensibility | Baseline
  Sensibility %
Assess the relevance of TPE for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Specificity | Baseline
  Specificity %
Assess the relevance of TPE for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Positive predictive values | Baseline
  Positive predictive values %
Assess the relevance of TPE for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Negative predictive values | Baseline
  Negative predictive values %
Assess the relevance of TPE for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Positive likelihood ratio | Baseline
  Positive likelihood ratio %
Assess the relevance of TPE for the etiological diagnosis of COPD decompensation in patients managed for ARD in the emergency department. Negative likelihood ratio | Baseline
  Negative likelihood ratio %
Assess the relevance of PTS for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Sensibility | Baseline
  Sensibility %
Assess the relevance of PTS for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Specificity | Baseline
  Specificity %
Assess the relevance of PTS for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Positive predictive values | Baseline
  Positive predictive values %
Assess the relevance of PTS for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Negative predictive values | Baseline
  Negative predictive values %
Assess the relevance of PTS for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Positive likelihood ratio | Baseline
  Positive likelihood ratio %
Assess the relevance of PTS for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Negative likelihood ratio | Baseline
  Negative likelihood ratio %
Assess the relevance of IPT for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Sensibility | Baseline
  Sensibility %
Assess the relevance of IPT for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Specificity | Baseline
  Specificity %
Assess the relevance of IPT for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Positive predictive values | Baseline
  Positive predictive values %
Assess the relevance of IPT for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Negative predictive values | Baseline
  Negative predictive values %
Assess the relevance of IPT for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Positive likelihood ratio | Baseline
  Positive likelihood ratio %
Assess the relevance of IPT for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Negative likelihood ratio | Baseline
  Negative likelihood ratio %
Assess the relevance of TPE for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Sensibility | Baseline
  Sensibility %
Assess the relevance of TPE for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Specificity | Baseline
  Specificity %
Assess the relevance of TPE for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Positive predictive values | Baseline
  Positive predictive values %
Assess the relevance of TPE for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Negative predictive values | Baseline
  Negative predictive values %
Assess the relevance of TPE for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Positive likelihood ratio | Baseline
  Positive likelihood ratio %
Assess the relevance of TPE for the etiologic diagnosis of PAO in patients managed for ARD in the emergency department; Negative likelihood ratio | Baseline
  Negative likelihood ratio %
Visually analyze the shape of the Diaphragmatic curves (DC) of patients seen for ARD in the emergency department and whose cause is mixed (association of at least two causes). | Baseline
  Descriptive analysis of curve shapes
Assessing the relevance of IPT for the etiological diagnosis of pneumopathy in patients managed for ARD in the emergency department. Positive predictive values | Baseline
  Positive predictive values %

CONTACTS AND LOCATIONS:
Overall Officials: DINO TIKVESA, MD, Principal Investigator — University Hospital, Montpellier
Locations (2):
- France (2):
  - University Hospital of Nîmes, Nîmes, Gard
  - University Hospital of Montpellier, Montpellier, Hérault

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jouneau S, Dres M, Guerder A, Bele N, Bellocq A, Bernady A, Berne G, Bourdin A, Brinchault G, Burgel PR, Carlier N, Chabot F, Chavaillon JM, Cittee J, Claessens YE, Delclaux B, Deslee G, Ferre A, Gacouin A, Girault C, Ghasarossian C, Gouilly P, Gut-Gobert C, Gonzalez-Bermejo J, Jebrak G, Le Guillou F, Leveiller G, Lorenzo A, Mal H, Molinari N, Morel H, Morel V, Noel F, Pegliasco H, Perotin JM, Piquet J, Pontier S, Rabbat A, Revest M, Reychler G, Stelianides S, Surpas P, Tattevin P, Roche N. Management of acute exacerbations of chronic obstructive pulmonary disease (COPD). Guidelines from the Societe de pneumologie de langue francaise (summary). Rev Mal Respir. 2017 Apr;34(4):282-322. doi: 10.1016/j.rmr.2017.03.034. Epub 2017 May 25. PMID 28552256
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; ESC Committee for Practice Guidelines. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012 Jul;33(14):1787-847. doi: 10.1093/eurheartj/ehs104. Epub 2012 May 19. No abstract available. PMID 22611136
- [Background] Abdallah S, Pihan F, Vandroux D. Échographie diaphragmatique : applications au-delà du sevrage de la ventilation. Le Praticien en Anesthésie Réanimation. 1 sept 2023;27(4):205-11.
- [Background] Jung B, Guillon A, pour la Commission de la recherche translationnelle de la SRLF. Échographie du diaphragme en réanimation. Schnell D, Charles PE, éditeurs. Méd Intensive Réa. janv 2019;28(1):60-3